CLINICAL TRIAL: NCT03252652
Title: Standardization of Normal Parameters of Cranial Vessels by Using Extra and Trans Cranial Vascular Duplex Among Egyptian Population
Brief Title: Normal Parameters of Cranial Vessels Using Cranial Vascular Duplex Among Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohammed Hamdy Ghazally, principle investigator, Assiut University
Other Study IDs: SNPCUETCDE
Record Dates: First submitted 2017-08-08; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Atherosclerosis; Atheroma of Cerebral Arteries; Atheroma; Carotid Artery; Atheroma; Cerebral
Keywords: Cranial vessels; Normal parameters; Carotid Duplex; Egyptian
MeSH Terms: conditions — Atherosclerosis; Carotid Artery Diseases; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: vascular duplex ultrasound imaging — Duplex ultrasound is a non-invasive evaluation of blood flow through cranial arteries and veins.

SUMMARY:
the study will be carried out to standardize normal parameters of vascular duplex ultrasound of the cranial vessels in the Egyptian population.

DETAILED DESCRIPTION:
Atherosclerosis is a major cause of ischemic stroke and a significant proportion of strokes are thromboembolic in nature, arising from atherosclerotic plaques. Several studies have reported racial differences in the severity and distribution of carotid atherosclerosis. In the United States and Western communities, Extra-cranial carotid artery disease was estimated to be responsible for 20-30% of strokes. Little is known about the prevalence and distribution of carotid disease among the populations in the developing countries.

Vascular duplex ultrasound is a useful, cheap and available diagnostic tool for assessing cranial vascular disease. Duplex ultrasound can be highly reliable with proper technique, without the risk of radiation in other imaging modalities, is well tolerated by all patients including those who are claustrophobic in MRI machines, and has much less risks compared to conventional angiography studies.

Although vascular duplex has been used for years yet there is little researches had been done on normal population in the developing countries to collect results and compare it to the parameters that was collected and reviewed in the western developed populations.

The parameters that would be used in this study include both the data collected by static and dynamic duplex scan which are the intimal-medial thickness, the vessels' diameter, peak flow velocity and peak flow volume both systolic and diastolic for either extra- or intra-cranial vessels.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects between 20-40 years

Exclusion Criteria:

* Diabetic patients, hypertensive patients, any evidence of vascular disease either peripheral or central, subjects refusing to participate

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Normal intimal-medial thickness measured in millimeter | 24 months
  Estimation of the intimal-medial thickness for cranial vessels.
Normal vessels' diameter measured in millimeter | 24 months
  Estimation of the vessels' diameter
Normal peak flow velocity measured in cm/sec | 24 months
  peak flow velocity both systolic and diastolic for cranial vessels
Normal indices | 24 months
  pulsatility index and resistance index for cranial vessels

SECONDARY OUTCOMES:
Early detection of subjects at risk of atherosclerosis | 24 months
  detection of subjects with early atherosclerotic changes for further management

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa H Ghazally, MBChB, Principal Investigator — Assiut University

REFERENCES:
- [Background] Yadav JS, Wholey MH, Kuntz RE, Fayad P, Katzen BT, Mishkel GJ, Bajwa TK, Whitlow P, Strickman NE, Jaff MR, Popma JJ, Snead DB, Cutlip DE, Firth BG, Ouriel K; Stenting and Angioplasty with Protection in Patients at High Risk for Endarterectomy Investigators. Protected carotid-artery stenting versus endarterectomy in high-risk patients. N Engl J Med. 2004 Oct 7;351(15):1493-501. doi: 10.1056/NEJMoa040127. PMID 15470212
- [Background] Grau AJ, Weimar C, Buggle F, Heinrich A, Goertler M, Neumaier S, Glahn J, Brandt T, Hacke W, Diener HC. Risk factors, outcome, and treatment in subtypes of ischemic stroke: the German stroke data bank. Stroke. 2001 Nov;32(11):2559-66. doi: 10.1161/hs1101.098524. PMID 11692017
- [Background] Timsit SG, Sacco RL, Mohr JP, Foulkes MA, Tatemichi TK, Wolf PA, Price TR, Hier DB. Early clinical differentiation of cerebral infarction from severe atherosclerotic stenosis and cardioembolism. Stroke. 1992 Apr;23(4):486-91. doi: 10.1161/01.str.23.4.486. PMID 1561677
- [Background] Svicero DJ, Doiche DP, Mamprim MJ, Heckler MC, Amorim RM. Ultrasound evaluation of common carotid artery blood flow in the Labrador retriever. BMC Vet Res. 2013 Oct 7;9:195. doi: 10.1186/1746-6148-9-195. PMID 24094043